CLINICAL TRIAL: NCT01849328
Title: Testing Spectrosense EVA System for Detection of Breast Cancer by Analyzing Volatile Organic Compounds (VOCs) in Exhaled Air
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Rauscher, Gregory E., M.D. PA (Individual)
Responsible Party: Sponsor
Other Study IDs: E-13-492
Record Dates: First submitted 2013-05-03; First posted 2013-05-08 (Estimated); Last update posted 2013-11-19 (Estimated); Status verified 2013-11

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Breast Cancer
- Healthy

SUMMARY:
Volatile Organic Compounds (VOC) in human breath are captured and analyzed by the Spectrosense EVA system, which is combination of a gas chromatography (GC) and software algorithm. The objective is to obtain a set or sets of VOC bio-markers that will provide the best discrimination between Breast Cancer sick population and healthy population. The gold standard for identifying sick/healthy population is biopsy proven breast cancer.

ELIGIBILITY:
Breast Cancer group:

Inclusion Criteria:

* Age from 18 years old
* Breast cancer positive biopsy
* Before any treatment
* Signed Informed Patient Consent

Exclusion Criteria:

* Age under 18 years old
* Neoadjovant treatment
* Post surgery for breast cancer
* A history of any other cancer type, except skin cancer that is not melanoma

Healthy group:

Inclusion Criteria:

* Healthy women
* No history of Breast cancer
* Signed Informed Patient Consent

Exclusion Criteria:

* History of Breast cancer
* Breast cancer background in the family
* A history of any other cancer type, except skin cancer that is not melanoma

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Women with breast cancer, biopsy confirmed, ages above 18. vs. Healthy women without breast cancer.
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2013-05; Primary Completion 2014-05 (Estimated)

PRIMARY OUTCOMES:
Obtaining a set or sets of VOC bio-markers that will provide the best discrimination between Breast Cancer sick population and healthy population. breast cancer. | Upon enrollment.

CONTACTS AND LOCATIONS:
Locations (1):
- Englewood Hospital and Medical Center, Englewood, New Jersey, United States